CLINICAL TRIAL: NCT01046331
Title: Novel Influenza A (H1N1) Surveillance Registry
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Andrea Harabin, National Heart, Lung, and Blood Institute (NHLBI)
Other Study IDs: 688; N01HR056179 (NIH); HSN268200536179C (Other Grant/Funding Number: NIH Contract Number)
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2010-11

CONDITIONS: Novel Influenza A; H1N1; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adult H1N1: Patients admitted to adult ICU with confirmed or suspected H1N1 Influence infection
- Pediatric H1N1: Patients admitted to pediatric ICU with confirmed or suspected H1N1 Influenza infection

SUMMARY:
The demographic characteristics, clinical features, course, and outcomes of severe H1N1 influenza infection requiring intensive care have not been defined rigorously and systematically. While the majority of patients in early reports of critically ill novel influenza A (H1N1) have respiratory involvement, up to 10-20% may present with non-respiratory organ failures, such as shock, seizures, or acute renal failure. The burden of disease and resource utilization of these patients remains largely unknown. The purpose of this surveillance registry is to characterize the demographics, clinical features, outcomes, and resource utilization of patients with H1N1 influenza infection who require intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Admission to an intensive care unit at a participating site with confirmed or suspected Novel H1N1 Influenza infection

Exclusion Criteria:

* Influenza-like illness due to non-influenza disease and negative testing for influenza

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects admitted to adult or pediatric ICUs with suspected or confirmed Novel H1N1 Influenza infection.
Sampling Method: Non-Probability Sample
Enrollment: 894 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B. Taylor Thompson, MD, Principal Investigator — Massachusetts General Hospital; Adrienne G Randolph, MD, MSc, Principal Investigator — Boston Children's Hospital; Todd W Rice, MD, MSc, Principal Investigator — Vanderbilt University
Locations (86):
- United States (86):
  - Alaska Native Medical Center, Anchorage, Alaska
  - The Children's Hospital at Providence, Anchorage, Alaska
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hiospital, Little Rock, Arkansas
  - University of San Francisco-Fresno Medical Center, Fresno, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California, Davis Medical Center, Sacramento, California
  - UCSF Children's Medical Center, San Francisco, California
  - UCSF-Moffitt Hospital, San Francisco, California
  - UCSF-San Francisco General Hospital, San Francisco, California
  - University of California, San Francisco (UCSF)-Moffitt Hospital, San Francisco, California
  - Denver's Children Hospital, Aurora, Colorado
  - Centura St. Anthony Central Hospital, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale-New Haven Children's Hospital, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic at Jacksonville, Jacksonville, Florida
  - Holt'z Children's Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Kapi'olani Center for Women and Children, Honolulu, Hawaii
  - Children's Memorial Hospital, Chicago, Illinois
  - Kosair Children's Hospital, Louisville, Kentucky
  - Earl K. Long Medical Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Medical Center of Louisiana, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Union Memorial Hospital, Baltimore, Maryland
  - University of Maryland Shock Trauma Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota Children's Hospital, Minneapolis, Minnesota
  - Rochester Methodist Hospital, Rochester, Minnesota
  - St. Mary's Hospital, Mayo Clinic, Rochester, Minnesota
  - SSM Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Nebraska, Omaha, Nebraska
  - Darthmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Rochester Medical Center, Rocherster, New York
  - Children's Hospital of Montefiore, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Children's Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Durham Regional Medical Center, Durham, North Carolina
  - Moses Cone Health System, Greensboro, North Carolina
  - Wesley Long Community Hospital, Greensboro, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Nationwide Children' Hospital, Columbus, Ohio
  - Children's Hospital at St. Francis, Tulsa, Oklahoma
  - Doernbecher Children's Hospital, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe Carell Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - University of Texas Southwestern Children's Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Virginia Children's Medical Center, Charlottesville, Virginia
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Providence Hospital, Everett, Washington
  - Harborview Medical Center, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Related Info — http://www.ardsnet.org
- Available data/document: Individual Participant Data Set: H1N1 — http://biolincc.nhlbi.nih.gov/studies/h1n1/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/h1n1/